CLINICAL TRIAL: NCT01567033
Title: Translating a Weight Loss Intervention Through a National Home Visiting Program
Brief Title: Healthy Eating and Active Living Taught at Home
Acronym: HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201103147
Record Dates: First submitted 2012-03-14; First posted 2012-03-30 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Diabetes; Obesity
Keywords: Diabetes; Obesity; Home visiting
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Intervention participants received HEALTH, which embedded a lifestyle intervention derived from DPP within the standard PAT curriculum
  Interventions: Behavioral: PAT Curriculum + Health Information

INTERVENTIONS:
Behavioral: PAT Curriculum + Health Information — Participants in the intervention group will receive the standard PAT curriculum plus information about healthy eating and an active lifestyle. This curriculum will be taught during up to 36 home visits in two years. Months 1-3 the visits are weekly; months 4-6 visits are biweekly; months 7-24 visits are monthly

SUMMARY:
The purpose of this research study is to evaluate two different Parents as Teachers curriculums taught by parent educators, during home visits. The control curriculum includes only the standard PAT lessons; the intervention curriculum includes the standard PAT lessons plus additional information about how families can live healthy and active lives while reaching a healthy weight. The investigators hypothesize the intervention lessons will change the way people eat and/or their activity level.

DETAILED DESCRIPTION:
The primary aim is to test Healthy Eating & Active Living Taught at Home (HEALTH), which adapts and integrates the Diabetes Prevention Program lifestyle intervention within Parents As Teachers (PAT), a national home visiting program on which many high needs populations rely for parent-child information and services. Specific aims 1 and 2 will evaluate the impact of HEALTH on lifestyle behaviors and weight of obese mothers and their overweight/obese preschool child across multiple PAT regions. Specific aims 3 and 4 will address elements of external validity through evaluation of factors that impact the uptake of HEALTH within the PAT organization.

Specific aim 1. Using a group randomized, nested cohort design, evaluate the impact of HEALTH on obese women (BMI 30-45 kg/m2; age 18-45 y old) randomized to either control regions receiving the standard PAT program, or intervention regions receiving HEALTH.

Hypothesis 1.1 The primary hypothesis is at the conclusion of the study, when compared to the control group, participants in HEALTH will achieve a 7% weight loss at 12 months and maintain a 5% weight loss at 24 months, which will be at least two-fold greater than that achieved in the control group.

The secondary hypotheses are that at the conclusion of the study, when compared to the control group, participants in HEALTH will significantly:

Hypothesis 1.2 Improve clinical outcomes of waist circumference and systolic and diastolic blood pressure; Hypothesis 1.3 Improve knowledge of evidence-based lifestyle behaviors and quality of life; Hypothesis 1.4 Decrease caloric intake Hypothesis 1.5 Increase moderate intensity walking.

Specific aim 2. The secondary aim is to determine whether improvements in 'mother to child' behaviors of HEALTH participants will explain all or part of changes in the weight trajectory of the participant's overweight (>85th percentile) or obese (>95th percentile) preschool child. The hypotheses are that at the conclusion of the study, when compared to the control group:

Hypothesis 2.1 There will be a significantly greater proportion of participants in the HEALTH group who improve child feeding practices with their preschool child; Hypothesis 2.2 There will be a significantly greater proportion of preschool children in the HEALTH group who maintain or reduce their weight as measured by BMI Z-score.

Specific aim 3. The aim is to assess and provide information on the external validity of HEALTH to enhance research translation (e.g. reach and representativeness, program implementation or adaptation, decision making outcomes, and maintenance or institutionalization).

Question 3.1 Are HEALTH adopters representative of control PAT participants and parent educators? Question 3.2 Are HEALTH parent educators effectively trained to deliver the intervention? Question 3.3 Is HEALTH implemented as designed or adapted for content, consistency, or intensity? Question 3.4 Is HEALTH maintained as an institutionalized component of PAT practice? Specific aim 4. The aim is to determine the cost-utility of HEALTH in decreasing obesity and risk for diabetes from two perspectives: the service provider and state health agencies.

Question 4.1 Is the implementation and maintenance of HEALTH effective from a cost-utility perspective for the participants enrolled in the program and the agencies considering implementing these programs? Question 4.2 Is HEALTH effective in improving health quality, from the perspective of state agencies considering funding decisions for this and similar programs?

ELIGIBILITY:
Inclusion Criteria:

* female, obese (BMI 30 -45 kg/m2),have at least one overweight or obese preschool child (>60th percentile) living in the home, plan to continue in the PAT program for two years, and able to give informed consent to participate in HEALTH.

Exclusion Criteria:

* current pregnancy or plan to become pregnant in the next 24 months, inability to speak English, current enrollment in any weight loss program, a diagnosis and/or undergoing treatment for diabetes, cardiovascular disease, or eating disorders, or inability to exercise or engage in a walking program.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 460 (Actual)
Dates: Start 2012-04-26 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Change in BMI from baseline to 24 months
  Body mass index (BMI) will be used to classify participants as "obese". The investigators will calculate the BMI from weight and height measurements. Participants weight measurement will be obtained using a calibrated scale placed on a solid flat surface. The screener will record the weight in pounds. Height measurement will be the maximum vertical height measured using a stadiometer on a solid flat surface with a fixed vertical backboard and an adjustable headpiece or an approved portable stadiometer on a solid flat surface with an adjustable headpiece.

SECONDARY OUTCOMES:
Waist Circumference | Change in waist circumference from baseline to 24 months
  Waist circumference will be used to estimate abdominal adiposity which is associated with risk of Type 2 diabetes.
Blood Pressure | Change in blood pressure from baseline to 24 months
  In accordance with American Heart Association guidelines, we will follow the recommendations and protocol for blood pressure measurement.
Survey | Changes in surveys from baseline to 24 months
  Survey includes: dietary screener, International Physical Activity Questionnaire, SF-12 to assess quality of life, a knowledge test to reflect the HEALTH intervention, questions asking about lifestyle patterns, environmental questions, sleep, Preschooler Feeding Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Debra Haire Joshu, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Tabak RG, Morshed AB, Schwarz CD, Haire-Joshu D. Impact of a Healthy Weight Intervention Embedded Within a National Home Visiting Program on the Home Food Environment. Front Public Health. 2018 Jun 26;6:178. doi: 10.3389/fpubh.2018.00178. eCollection 2018. PMID 29998092
- [Derived] Haire-Joshu D, Schwarz CD, Steger-May K, Lapka C, Schechtman K, Brownson RC, Tabak RG. A Randomized Trial of Weight Change in a National Home Visiting Program. Am J Prev Med. 2018 Mar;54(3):341-351. doi: 10.1016/j.amepre.2017.12.012. PMID 29455756